CLINICAL TRIAL: NCT01632748
Title: Validation Study in Healthy Female Volunteers: A Comparison of Two Neurotech Vital Devices Set up to Provide Different Types of Electrical Stimulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Medical Research, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single
Other Study IDs: BMR-12-1004
Record Dates: First submitted 2012-06-29; First posted 2012-07-03 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-06

CONDITIONS: Healthy Female Volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified Neurotech Vital Device (Experimental): Checking to observe stimulation delivered using this device
  Interventions: Device: Modified Neurotech Vital Device
- Neurotech Vital Device (Active Comparator): Checking to see if stimulation observed using this device
  Interventions: Device: Neurotech Vital Device

INTERVENTIONS:
Device: Neurotech Vital Device — 5 minute treatment
  Other Names: Modified Neurotech Vital Device
  Arms: Neurotech Vital Device
Device: Modified Neurotech Vital Device — 5 minute stimulation
  Arms: Modified Neurotech Vital Device

SUMMARY:
This research is being carried out in order to compare two alternative versions of the Neurotech Vital Devices which have been set up to provide two different types of stimulation. Both these devices will be fully functioning devices and the investigators want to collect information on your perception of the two alternative modes. The patient will be asked to provide feedback on both devices which will look identical. The patient will not be told in which order the units were given to them until the completion of your visit.

DETAILED DESCRIPTION:
The Neurotech Vital Device is connected to a series of conductive hydrogel electrodes strategically positioned in and around the pelvic area of the user. The electrode positions and current pathways deliver therapeutic stimulation to the pelvic floor muscles resulting in repeated contraction of the intended muscle group. Pilot study data has shown this novel approach to produce extremely favorable adaptation and improvement in patient's symptoms following intervention. In order to capture the intended electrode position a stand-alone garment that will allow the end user to re-position electrodes on multiple re-applications is required. The Neurotech Vital Device garment is CE Marked as a Class IIa medical device and it is CE Marked, as part of the Neurotech Vital Device, in line with Medical Device Directive 93/42/EC as amended by 2007/47/EC. The Neurotech Vital Device garment is not cleared by the FDA through the 510 (k) pre-market notification process in the USA but would be considered a Class II device as part of the Neurotech Vital Device.

The purpose of this validation study is to establish the suitability of the Neurotech Vital device in which the treatment stimulation parameters have been markedly attenuated (defined as 'modified Neurotech Vital device') prior to its use as one of the treatments in a randomised, controlled, double-blind study to be conducted in patients with stress urinary incontinence in Germany (Study No: BMR-11-1002).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are female and at least 18 years of age.
* Subjects who, in the opinion of the Investigator, are deemed healthy.
* Subjects who are able to give voluntary, written informed consent to participate in this study and from whom consent has been obtained.
* Subjects who are able to understand this study and are willing to complete all the study assessments.

Exclusion Criteria:

* Subjects who have a physical condition that would make them unable to perform the study procedures.
* Subjects with a history of any chronic respiratory condition (ie emphysema, chronic obstructive pulmonary disease).
* Subjects with a history of an underlying neurological condition.
* Subjects with a history of low back pain involving the spinal nerve root.
* Subjects with a blood clotting disorder or who are taking anti-coagulant medications.
* Subjects who have previously had any uro-gynaecological related surgery excluding hysterectomy.
* Subjects with a clinical diagnosis of prolapse greater than Stage 2.
* Subjects who are pregnant or could be pregnant.
* Subjects who are less than 6 months post-partum or who are lactating.
* Subjects who have any intra-uterine devices or metal implants in the pelvic area, including hip and lumbar spine.
* Subjects with pelvic pain or fibromyalgia or paravaginal defect.
* Subjects with an active implanted medical device (ie pacemaker, pump etc).
* Subjects with a history of heart disease or stroke.
* Subjects with a known cancer.
* Subjects with an injury or disability affecting any part of their body which will be in contact with the garment.
* Subjects who are currently involved in any injury litigation claims.
* Subjects who have been committed to an institution by virtue of an order issued either by the courts or by an authority.
* Subjects who have participated in a clinical study in the last 3 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The primary objective of this validation study is to verify that the Modified Neurotech Vital Device does not elicit a pelvic floor contraction compared to the Neurotech Vital Device. | Day1
  The primary endpoint of the study is to demonstrate that no volunteers elicit a contraction of the pelvic floor muscle with the Modified Neurotech Vital Device and that all the volunteers elicit a contraction of the pelvic floor muscle with the Neurotech Vital Device. Contraction of the pelvic floor muscles will be assessed by using sonographic/real time ultrasound imaging/recording (mean of three measurements of pelvic floor displacement achieved during maximum threshold intensity electrical stimulation).

SECONDARY OUTCOMES:
The secondary objective of this validation study is to verify that the Modified Neurotech Vital Device is perceived by the volunteers as a valid treatment option in terms of sensation. | Day1
  Subjects will also be asked to complete a feedback questionnaire on the use of the Modified Neurotech Vital Device to verify that it is perceived as a valid treatment option.

CONTACTS AND LOCATIONS:
Locations (1):
- North Georgia College and State University, Dahlonega, Georgia, United States